CLINICAL TRIAL: NCT05547763
Title: THE EFFICACY OF RESORBABLE PLATES VERSUS TITANIUM PLATES IN TERMS OF STABILITY AMONG PATIENTS WITH MANDIBULAR FRACTURES: A RANDOMIZED CONTROLLED TRIAL.
Brief Title: THE EFFICACY OF RESORBABLE PLATES VERSUS TITANIUM PLATES IN TERMS OF STABILITY IN MANDIBULAR FRACTURES.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUHS/BASR/2019/-515
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Comparison of Resorbable Plates With Titanium Plates
Keywords: Resorbable plates,titanium plates,stability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resorbable plates, test group (Experimental): after a surgical procedure under general anesthesia , resorbable plates will be placed on the fracture site of the mandibule in 20 patients out of 40 total sample size and will be compared with the titanium plates in the control group
  Interventions: Procedure: surgically mandible will be exposed to reduced the fracture anatomically and then fixated with either resorbable or the titanium plates
- titatnium plates, control group (Experimental): after a surgical procedure under general anesthesia , titanium plates will be placed on the fracturte site in the mandible in 20 patients out of 40 total sample size and will be compared to the test group containing resorbable plates
  Interventions: Procedure: surgically mandible will be exposed to reduced the fracture anatomically and then fixated with either resorbable or the titanium plates

INTERVENTIONS:
Procedure: surgically mandible will be exposed to reduced the fracture anatomically and then fixated with either resorbable or the titanium plates — under general anesthesia , fracture site of the mandible will be exposed and fracture will be reduced anatomically and held together by either resorbable or titanium plates and then the incsion site will be closed with vicryl sutures and patient will be observed on the follow ups clinically and radiographically for the fracture reduction and stability of the fractures with resorbable plates as compared to the titanium plates.

SUMMARY:
Objective To compare the efficacy of resorbable plates against titanium plates to determine the fixation stability in reducing mandibular fractures

Method:

Subjects will be recruited and divided into two groups by random allocation. Consents will be obtained and fracture sites will be examined clinically and radiographically. Control group will receive titanium plates and test group will receive resorbable plates. The patients will be recalled immediately at first postop day then at the end of the first month , second month and the third month.They will be evaluated for the reduction of the fractures.

DETAILED DESCRIPTION:
Study design:

randomized controlled trial

Study Setting:

The study will be carried out at the Department Of Oral and maxillofacial Surgery in Dow University of Health Sciences and Civil Hospital Karachi

Study Population:

Samples will be recruited by setting the following criteria:

Inclusion Criteria:

* Age group-18 years and above
* Symphysis and body fractures.
* Non-infected fracture site

Exclusion Criteria:

* Condylar fracture
* Comminuted fractures
* Patients with systemic bone diseases
* Gunshot wounds
* Pan-facial trauma
* Infected wounds

Sample Size:

Total 40 patients will be carried out (20 in treatment & 20 in control group). Using PASS version 11, two sample proportions with 95% confidence interval, 90% power of the test, 100% proportion of union of the fracture in resorbable fixation (treatment group) and 99% in titanium (control group),calculated sample size is 35 in each group keeping the population at approximately 120 patients in six months, calculated sample size is 70 patients.(18) But due to the budget constraints treatment group (resorbable fixation) will contain 20 patients and control group (titanium) will contain 20 patients

Sampling Technique:

Consecutive Sampling

Data Collection Procedure:

Data will be collected from the patients after receiving informed consent. Baseline demographic variable will be recorded using a predesigned questionnaire. Patients will be allocated to either resorbable or titanium plate group through random allocation [through lottery method]. Assessment will be done clinically and radiographically on CBCT scan (available at Dow International Dental College) First follow up assessment will be done immediately post op. Further assessments will be done at the completion of 2nd month and and then the 3rd month.

Statistical Analyses:

Data will be entered and analyzed using SPSS v 22. Mean and standard deviation will be calculated for all continuous variables, whereas frequencies and percentages will be calculated for all categorical variables. Efficacy of the intervention group will be assessed using chi-squared test.

Study Variables

Independent Variables:

Interventions: Titanium or Resorbable plates

Dependent Variables Fixation stability

Co-variates:

Age, Gender, Fracture site

ELIGIBILITY:
Inclusion Criteria:

* • Age group-18 years and above

  * Symphysis and body fractures.
  * Non-infected fracture site

Exclusion Criteria:

* • Condylar fracture

  * Comminuted fractures
  * Patients with systemic bone diseases
  * Gunshot wounds
  * Pan-facial trauma
  * Infected wounds

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-11-09 (Estimated); Study Completion 2022-11-09 (Estimated)

PRIMARY OUTCOMES:
bone union | 3 months
  union of the fractured bone will be observed radiographically at the end of the first ,second and the third month by a cone beam computed tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No